CLINICAL TRIAL: NCT00103259
Title: Phase II Two Arm Trial of the Proteasome Inhibitor, PS-341 (Velcade TM) in Combination With Irinotecan or PS-341 Alone Followed by the Addition of Irinotecan at Time of Progression in Patients With Locally Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck (SCCHN)
Brief Title: Bortezomib With or Without Irinotecan in Treating Patients With Locally Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NCI-2012-02953; NCI-2012-02953 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); E1304 (Other: Eastern Cooperative Oncology Group); E1304 (Other: CTEP); U10CA021115 (NIH); NCT00695721 (obsolete NCT alias)
Record Dates: First submitted 2005-02-07; First posted 2005-02-08 (Estimated); Results first posted 2012-12-27 (Estimated); Last update posted 2014-05-23 (Estimated); Status verified 2012-12

CONDITIONS: Recurrent Squamous Cell Carcinoma of the Hypopharynx; Recurrent Squamous Cell Carcinoma of the Larynx; Recurrent Squamous Cell Carcinoma of the Lip and Oral Cavity; Recurrent Squamous Cell Carcinoma of the Nasopharynx; Recurrent Squamous Cell Carcinoma of the Oropharynx; Recurrent Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Recurrent Verrucous Carcinoma of the Larynx; Recurrent Verrucous Carcinoma of the Oral Cavity; Stage IV Squamous Cell Carcinoma of the Hypopharynx; Stage IV Squamous Cell Carcinoma of the Larynx; Stage IV Squamous Cell Carcinoma of the Nasopharynx; Stage IV Verrucous Carcinoma of the Larynx; Stage IVA Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IVA Squamous Cell Carcinoma of the Oropharynx; Stage IVA Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage IVA Verrucous Carcinoma of the Oral Cavity; Stage IVB Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IVB Squamous Cell Carcinoma of the Oropharynx; Stage IVB Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage IVB Verrucous Carcinoma of the Oral Cavity; Stage IVC Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IVC Squamous Cell Carcinoma of the Oropharynx; Stage IVC Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage IVC Verrucous Carcinoma of the Oral Cavity; Tongue Cancer
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Tongue Neoplasms | interventions — Bortezomib; Irinotecan

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Arm I (bortezomib, irinotecan hydrochloride) (Experimental): Patients receive bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11 and irinotecan IV over 90 minutes on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity
  Interventions: Drug: bortezomib; Drug: irinotecan hydrochloride; Other: laboratory biomarker analysis
- Arm II (bortezomib) (Experimental): Patients receive bortezomib as in arm I. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Upon disease progression, patients may cross over to arm I.
  Interventions: Drug: bortezomib; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: bortezomib — Given IV
  Other Names: LDP 341; MLN341; VELCADE
Drug: irinotecan hydrochloride — Given IV
  Other Names: Campto; Camptosar; CPT-11; irinotecan; U-101440E
  Arms: Arm I (bortezomib, irinotecan hydrochloride)
Other: laboratory biomarker analysis — Optional correlative studies

SUMMARY:
This randomized phase II trial is studying bortezomib and irinotecan to see how well they work compared to bortezomib alone in treating patients with locally recurrent or metastatic squamous cell carcinoma of the head and neck. Bortezomib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as irinotecan, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving bortezomib together with irinotecan may kill more tumor cells. It is not yet known whether giving bortezomib together with irinotecan is more effective than bortezomib alone in treating head and neck cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the activity of combination of PS-341 (bortezomib) and irinotecan in patients with locally advanced, recurrent or metastatic squamous cell carcinoma of the head and neck (SCCHN) and the response rate of single agent PS-341 (followed by irinotecan at time of progression).

SECONDARY OBJECTIVES:

I. To continue exploring the toxicity of PS-341 alone and the combination of PS-341 and irinotecan in this patient population.

II. To evaluate time to progression, overall survival and response to irinotecan and PS-341 when given after PS-341 alone.

III. To evaluate the relationship between pre-treatment nuclear localization of NF-kB, and NF-kB regulated gene expression in tissue (Cyclin D1, IAP1, Bcl-XL, Topo I), and serum (IL-6, IL-8, GRO-1 and VEGF) and response.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

Arm I: Patients receive bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11 and irinotecan IV over 90 minutes on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Arm II: Patients receive bortezomib as in arm I. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Upon disease progression, patients may cross over to arm I.

Patients are followed every 3-6 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients may have had one (0-1) prior chemotherapy regimen for recurrent or metastatic SCCHN; chemotherapy for recurrent or metastatic disease must have been completed at least 4 weeks prior to study entry
* Patients must not have been previously treated with irinotecan or bortezomib

  * Patients must not be receiving radiation treatment
* Patients must have histologically confirmed squamous cell carcinoma of the head and neck
* Patients must have biopsy for histological confirmation of recurrent or metastatic disease if disease is now recurrent or metastatic after prior disease free-interval

  * NOTE: If patient has had a complete response (of any duration) but now has suspected recurrent disease (regardless of the time interval), the patient will need a biopsy for confirmation of SCCHN
* Disease must not be amenable to potentially curative local therapies or patient must have refused such options
* Patients must not have nasopharyngeal subtypes WHO II or III. Patients may have nasopharyngeal WHO I; salivary gland primaries are excluded from study SUBTYPES OF NASOPHARYNGEAL CARCINOMA (NPC) WHO type 1 - keratinizing SCC WHO type 2 - nonkeratinizing epidermoid carcinoma WHO type 3 - undifferentiated carcinoma
* Patients must have measurable disease

  * Baseline measurements and evaluations must be obtained within 4 weeks of registration to the study
  * Measurable disease limited to a pre-irradiated location must be biopsy proven to be squamous cell carcinoma
* Must have at least one objective measurable disease parameter; baseline measurements and evaluations must be obtained within 4 weeks of registration to the study; all areas of disease should be recorded and mapped out in order to assess response and uniformity of response to therapy

  * Radiographic findings are acceptable providing that clear-cut measurement can be made
  * Measurable disease limited to a pre-irradiated location must be biopsy-proven to be squamous cell carcinoma
* Patients must have ECOG performance status 0 or 1
* Patients must not have grade 2 or higher peripheral neuropathy within 2 weeks of study entry
* Leukocytes >= 3,000/uL
* Absolute neutrophil count >= 1,500/uL
* Platelets >= 100,000/uL
* Total bilirubin within normal institutional limits
* AST(SGOT) and ALT(SGPT) =< 2.5 x institutional upper limit of normal
* Creatinine within normal institutional limits OR
* Creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Patients must have had no prior invasive malignancy unless the disease-free interval is 5 years or more
* Women must not be pregnant or breast-feeding due to the fact that the teratogenic or abortifacient effects of PS-341are unknown; the effect of PS-341 on the nursing infant are also unknown; all females of childbearing potential must have a blood test or urine study within 2 weeks prior to registration to rule out pregnancy
* Women of childbearing potential and sexually active males must be strongly advised to use an accepted and effective method of contraception for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Patients with known brain metastases will be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* Patients must not have history of allergic reactions to PS-341 or allergic reaction attributed to compounds of similar chemical or biologic composition to PS-341 including boron or mannitol
* Patients must not have uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, unstable angina pectoris, or psychiatric illness/social situations that would limit compliance with study requirements
* ELIGIBILITY FOR RE-REGISTRATION TO ARM A (FOR ARM B PATIENTS AT THE TIME OF PROGRESSION

  * Patients must have ECOG performance status 0 or 1
  * Leukocytes >= 3,000/uL
  * Absolute neutrophil count >- 1,500/uL
  * Platelets >= 100,000/uL
  * Total bilirubin within normal institutional limits
  * AST(SGOT) and ALT(SGPT) =< 2.5 x institutional upper limit of normal
  * Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
  * Patients with known brain metastases will be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2005-07; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill Gilbert, Principal Investigator — Eastern Cooperative Oncology Group
Locations (1):
- Eastern Cooperative Oncology Group, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: E1304 was open to accrual on July 20, 2005 and was suspended on September 29, 2006. The trial was reactivated on October 18, 2006 with dose reduction for irinotecan. Arm I was closed with 27 patients after stage I. Arm B proceeded to the second stage of accrual without suspension and closed on September 24, 2008 after enrolling 44 patients.
Groups:
- Arm I (Bortezomib+Irinotecan): Patients receive bortezomib IV over 3-5 seconds on days 1, 4, 8, and 11 and irinotecan hydrochloride IV over 90 minutes on days 1 and 8. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
- Arm II (Bortezomib): Patients receive bortezomib (PS-341) 1.3 mg/m2 IV over 3-5 seconds twice weekly on days 1, 4, 8 and 11 followed by one week of rest. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Upon disease progression, patients may cross over to arm I (bortezomib + irinotecan).
Period: Overall Study
Arm/Group | Arm I (Bortezomib+Irinotecan) | Arm II (Bortezomib)
Started | 27 | 44
Eligible | 27 | 41
Treated | 23 | 41
Eligible and Treated | 23 | 38
Cross Over to the Other Arm | 0 | 11 (11 patients who progressed on bortezomib crossed over to Arm I. 10 of them were eligible)
Eligible Patients Who Cross Over | 0 | 10
Completed | 15 (Treatment continued until disease progression or intolerable toxicity.) | 32 (Treatment continued until disease progression or intolerable toxicity.This number is for stage I.)
Not Completed | 12 | 12
Not completed — Death | 3 | 2
Not completed — Withdrawal by Subject | 2 | 3
Not completed — alternative therapy | 1 | 0
Not completed — other (reasons were not specified) | 2 | 1
Not completed — ineligible/no protocol therapy | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Bortezomib+Irinotecan) | Arm II (Bortezomib) | Total
Number analyzed (Participants) | 23 | 38 | 61
Age, Continuous [Median (Full Range); unit: years] | 61 [36 to 85] | 61 [45 to 78] | 61 [36 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 19 | 33 | 52
Region of Enrollment [Number; unit: participants]
  United States | 23 | 38 | 61

OUTCOME MEASURES:

1. Primary Outcome: Response Rate on Step 1
Description: Tumor response was evaluated via Response Evaluation Criteria In Solid Tumors (RECIST) v1.0, and response rate was defined as the proportion of patients with a complete response or partial response among all eligible and treated patients. Complete response was defined as disappearance of all tumor lesions. Partial response was defined as at least a 30% decrease in the sum of the longest diameters of target lesions.
Time Frame: Tumor response was assessed every 2 cycles until progression or intolerable toxicity with maximum of 3 years
Population: 61 eligible and treated patients were included in the analysis
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (Bortezomib+Irinotecan) | Arm II (Bortezomib)
Number analyzed (Participants) | 23 | 38
percentage of participants | 13.1 [3.6 to 30.3] | 2.6 [0.4 to 22.1]

2. Secondary Outcome: Response Rate on Step 2
Description: as for outcome 1
Time Frame: Tumor response was assessed after every 2 cycles until progression or intolerable toxicity with maximum of 3 years
Population: 10 eligible and treated patients who progressed on bortezomib and crossed over to bortezomib and irinotecan arm were included in the analysis
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- Cross-over From Bortezomib to Combined Arm: Patients progressed on bortezomib in step 1 crossed over to the combination arm. Response rate is evaluated in these patients.
Arm/Group | Cross-over From Bortezomib to Combined Arm
Number analyzed (Participants) | 10
percentage of participants | 0 [0 to 25.9]

3. Secondary Outcome: Progression-free Survival on Step 1
Description: Progression-free survival was defined as time from registration to step 1 to disease recurrence or death from any cause, whichever occurred first. Disease progression was measured by Response Evaluation Criteria In Solid Tumors (RECIST) v1.0, and defined as at least a 20% increase in the sum of the longest diameters of target lesions.
Time Frame: Every 3 months for first 2 years from protocol entry, then every 6 months until 3 years from study entry
Population: 61 eligible and treated patients were included in the analysis
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Bortezomib+Irinotecan) | Arm II (Bortezomib)
Number analyzed (Participants) | 23 | 38
months | 1.6 [1.2 to 7.3] | 1.5 [1.4 to 2.7]

4. Secondary Outcome: Overall Survival on Step 1
Description: Overall survival was defined as time from registration on step 1 to death from any cause. It was evaluated in all 61 eligible and treated patients.
Time Frame: Survival was assessed every 3 month within 2 years and every 6 months betwen 2 and 3 years
Population: 61 eligible and treated patients were included in the analysis
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Bortezomib+Irinotecan) | Arm II (Bortezomib)
Number analyzed (Participants) | 23 | 38
months | 9.1 [2.3 to 12.5] | 7.3 [5.1 to 9.4]

ADVERSE EVENTS:
Time Frame: Toxicity is assessed at the end of each cycle (1 cycle = 21 days) and at the 30 days following the last dose of protocol drug, or until the initiation of subsequent treatment, whichever comes first.
Description: All patients who received protocol therapy were evaluated for toxicity, regardless of eligibility
Groups:
- Cross-over Patients: 11 patients crossed over to bortezomib + irinotecan after progressed on bortezomib single agent. Adverse events were reported for the 11 patients while receiving the combination therapy.
Arm/Group | Arm I (Bortezomib+Irinotecan) | Arm II (Bortezomib) | Cross-over Patients
Serious Adverse Events (participants affected / at risk) | 17/23 | 21/41 | 6/11
Other Adverse Events (participants affected / at risk) | 23/23 | 40/41 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Bortezomib+Irinotecan) (N=23) | Arm II (Bortezomib) (N=41) | Cross-over Patients (N=11)
Anemia (Blood and lymphatic system disorders) | 4 | 2 | 0
Leukopenia (Leukocytes decreased) (Investigations) | 5 | 1 | 2
Lymphopenia (Investigations) | 1 | 4 | 1
Neutropenia (Neutrophils decreased) (Investigations) | 4 | 1 | 1
Thrombocytopenia (Platelets decreased) (Investigations) | 4 | 1 | 1
Hypotension (Vascular disorders) | 2 | 2 | 0
Fatigue (General disorders) | 0 | 7 | 1
Fever w/o neutropenia (General disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0
Constitutional, other (General disorders) | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 3 | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 4 | 0 | 3
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 5 | 1 | 1
Nausea (Gastrointestinal disorders) | 3 | 0 | 0
Vomiting (Gastrointestinal disorders) | 4 | 0 | 0
Stomach, hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Infection w/ gr3-4 neut, lung (Infections and infestations) | 1 | 0 | 1
Infection w/ gr0-2 neut, lung (Infections and infestations) | 1 | 0 | 0
Infection w/ gr0-2 neut, trachea (Infections and infestations) | 0 | 1 | 0
Infection w/ unknown ANC foreign body (Infections and infestations) | 1 | 0 | 0
Infection w/ gr0-2 neut, blood (Infections and infestations) | 1 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Glomerular filtration rate decreased (Renal and urinary disorders) | 1 | 0 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 3 | 2 | 1
Hyponatremia (Metabolism and nutrition disorders) | 4 | 1 | 0
Non-neuropathic generalized weekness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 4 | 0
Neuropathy-sensory (Nervous system disorders) | 0 | 3 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Abdomen, pain (Gastrointestinal disorders) | 0 | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Vessel injury carotid (Injury, poisoning and procedural complications) | 1 | 0 | 0
Death, NOS (General disorders) | 1 | 0 | 0
Obstruction, small bowel NOS (Gastrointestinal disorders) | 0 | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Bortezomib+Irinotecan) (N=23) | Arm II (Bortezomib) (N=41) | Cross-over Patients (N=11)
Anemia (Blood and lymphatic system disorders) | 21 | 31 | 10
Leukopenia (Leukocytes decreased) (Investigations) | 12 | 5 | 5
Lymphopenia (Investigations) | 2 | 1 | 0
Neutropenia (Neutrophils decreased) (Investigations) | 6 | 1 | 3
Thrombocytopenia (Platelets decreased) (Investigations) | 12 | 14 | 7
Hematologic-other (Blood and lymphatic system disorders) | 2 | 2 | 0
Hypotension (Vascular disorders) | 2 | 4 | 2
Fatigue (General disorders) | 14 | 17 | 8
Fever w/o neutropenia (General disorders) | 3 | 2 | 0
Insomnia (Psychiatric disorders) | 2 | 3 | 2
Weight loss (Investigations) | 5 | 4 | 3
Constitutional, other (General disorders) | 4 | 5 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 3 | 2
Rash/desquamation (Skin and subcutaneous tissue disorders) | 3 | 1 | 1
Anorexia (Metabolism and nutrition disorders) | 4 | 9 | 5
Constipation (Gastrointestinal disorders) | 2 | 12 | 2
Dehydration (Metabolism and nutrition disorders) | 2 | 1 | 0
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 14 | 11 | 4
Dry mouth (Gastrointestinal disorders) | 0 | 4 | 2
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 1 | 3 | 1
Nausea (Gastrointestinal disorders) | 11 | 13 | 6
Taste disturbance (Gastrointestinal disorders) | 1 | 4 | 1
Vomiting (Gastrointestinal disorders) | 4 | 9 | 6
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 | 2 | 1
Alkaline phosphatase increased (Investigations) | 2 | 3 | 0
Alanine aminotransferase increased (ALT, SGPT) (Investigations) | 1 | 3 | 2
Aspartate aminotransferase increased (AST, SGOT) (Investigations) | 2 | 5 | 3
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Creatinine increased (Investigations) | 3 | 0 | 1
Hyperglycemia (Investigations) | 1 | 3 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 2 | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 4 | 0
Hypokalemia (Metabolism and nutrition disorders) | 6 | 3 | 1
Hyponatremia (Metabolism and nutrition disorders) | 8 | 10 | 7
Dizziness (Nervous system disorders) | 3 | 4 | 4
Anxiety (Psychiatric disorders) | 0 | 4 | 1
Neuropathy- sensory (Nervous system disorders) | 5 | 13 | 4
Vision blurred (Eye disorders) | 2 | 1 | 0
Abdomen, pain (Gastrointestinal disorders) | 2 | 2 | 1
Back, pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Neuropathic, pain (Nervous system disorders) | 0 | 3 | 0
Stomach, pain (Gastrointestinal disorders) | 2 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 1
Sweating (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Weight gain (Investigations) | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Wound, non-infectious (Injury, poisoning and procedural complications) | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal disorders (GI)-other (Gastrointestinal disorders) | 0 | 0 | 1
Infection Gr0-2 neut, upper airway (Infections and infestations) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1
Bone, pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Head/headache (Nervous system disorders) | 0 | 0 | 1
Muscle, pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Neck, pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Throat/pharynx/larynx, pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Urethra, pain (Renal and urinary disorders) | 0 | 0 | 1
Voice change/dysarthria (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Edema head and neck (General disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less